CLINICAL TRIAL: NCT02922894
Title: Treatment of Sleep Apnea in Patients With Cervical Spinal Cord Injury
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: John D. Dingell VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1607015110; CDMRP-SC150201 (Other: Congressionally Directed Medical Research Program Office)
Record Dates: First submitted 2016-09-23; First posted 2016-10-04 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Apnea; Spinal Cord Injury
MeSH Terms: conditions — Sleep Apnea Syndromes; Spinal Cord Injuries | interventions — Trazodone; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Acute episodic hypoxia (Experimental): To test development of ventilatory augmentation following episodic hypoxia, defined as increased Hypoxic Ventilatory Response (HVR) from early to late hypoxic exposure episodes.
  Interventions: Procedure: Acute episodic hypoxia; Procedure: Sham
- Supplemental oxygen (Experimental): To use supplemental oxygen to decrease peripheral chemoreceptor activity in patients with SCI and central SDB. In addition, perform a repeat evaluation after treatment with supplemental oxygen or sham O2 for 6 weeks to determine if correction of chronic intermittent hypoxia, which mitigates sensory LTF, results in decreased propensity to central apnea.
  Interventions: Procedure: Supplemental oxygen; Procedure: Sham
- Trazodone or placebo (Experimental): examine the effect of trazodone on breathing during sleep
  Interventions: Drug: Trazodone; Drug: Placebo

INTERVENTIONS:
Procedure: Acute episodic hypoxia — The subjects will undergo 30 minutes of baseline monitoring followed by 15 episodes of one minute of episodic hypoxia with supplemental CO2 to maintain isocapnia. This is followed by a 45 minute recovery period.
  Arms: Acute episodic hypoxia
Procedure: Supplemental oxygen — Supplemental oxygen therapy for 6 weeks
  Arms: Supplemental oxygen
Drug: Trazodone — 100mg before bedtime
  Arms: Trazodone or placebo
Drug: Placebo — One placebo pill before-bedtime
  Arms: Trazodone or placebo
Procedure: Sham — Room air will be administered instead of episodic hypoxia or supplemental oxygen..
  Arms: Acute episodic hypoxia; Supplemental oxygen

SUMMARY:
This study will investigate potential therapeutic approaches for sleep-disordered breathing (SDB) in patients with chronic cervical spine injury (>6 months post-injury).

DETAILED DESCRIPTION:
Patients with cervical spinal cord injury demonstrate central sleep disordered breathing manifesting as central sleep apnea or a periodic breathing pattern. Understanding the causes of central sleep apnea may be critically important to understanding upper airway obstruction in susceptible individuals, given the critical role of ventilatory motor output in maintaining upper airway patency as evidenced by upper airway narrowing or occlusion at the nadir of ventilator drive during periodic breathing. This study is likely to identify therapeutic strategies that could be tested in large clinical trials, with the ultimate goal of improving quality of life among patients with cervical SCI who also experience central sleep disordered breathing.

To this end the research proposal is aimed as follows:

Specific Aim 1: Test the hypothesis that patients with cervical SCI will demonstrate greater magnitude of long-term facilitation (LTF) following episodic hypoxia during sleep, compared to patients with thoracic Spinal cord injury. This aim will be accomplished by measuring the effect of acute episodic hypoxic ventilation and upper airway mechanics in both groups.

Specific Aim 2: Test the hypothesis that dampening peripheral chemoreceptor activity in patients with cervical SCI and central sleep disordered breathing (SDB) with supplemental oxygen will reduce central respiratory events and decrease respiratory variability during sleep. The aim will be accomplished by providing supplemental oxygen to participants with cervical SCI and central SDB.

Specific Aim 3: Test the hypothesis that administration of trazodone, in patients with cervical spinal cord injury and central SDB will decrease respiratory related arousals and central apnea index, and the propensity to develop central apnea, compared to placebo. To accomplish this aim, the investigators will test the acute effect of trazodone on respiratory related arousals and central sleep apnea, and the chronic effect on central apnea indices and the CO2 reserve.

The investigators will study subjects with SCI at T6 or above who are not on artificial ventilation. To characterize the sleep and breathing state of each subject, polysomnography and upper airway collapsibility will be measured at baseline. Then the following experiments will be conducted: an episodic hypoxia protocol vs normoxia will be used to determine whether cervical SCI will demonstrate greater magnitude of LTF. Experiments will be conducted to see whether dampening peripheral chemoreceptor activity in cervical SCI by giving supplemental oxygen will reduce the central respiratory events and reduce the breathing variability during sleep. A cross over experiment will be done to see whether administration of trazodone in patients with cervical SCI and central SDB decreases respiratory-related arousals and central apnea. The participant will be given the drug/placebo for one week then cross over after a 1 week wash out period to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adults between the ages of 18 - 89
2. chronic spinal cord injury patients (T6 and above), > 3 months since injury and not on mechanical ventilation, and have not received mechanical ventilation via tracheostomy in the past.

Exclusion Criteria:

1. subjects ≤ 17 yrs old
2. Pregnant and lactating females
3. History of head trauma that resulted in neurological symptoms or loss of consciousness
4. advanced heart, lung, metabolic, liver or chronic kidney disease.
5. severe obstructive or restrictive respiratory defect by PFTs or history of tracheostomy
6. extreme obesity defined for this protocol as BMI ≥ 40 kg/m2 (to avoid the effect of morbid obesity on ventilation).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Tidal Volume | 1 Week
  Change in tidal volume from baseline to recovery period.
Change in CO2 reserve (Delta-PETCO2-AT) | 1 Week
  CO2 reserve is the requisite change to induce central apnea is referred to as the CO2 reserve, which can be positive or negative
Change in Apnea Hypopnea Index (AHI) | 1 week
  AHI is used to indicate the severity of sleep apnea.
Change in hypocapnic apneic threshold | 1 week
  The nadir pressure in the upper airway (supra-glotic pressure) prior to the occurrence of an arousal. This is a physiological parameter.

CONTACTS AND LOCATIONS:
Overall Officials: M Safwan Badr, M.D., Principal Investigator — John D. Dingell VA Medical Center
Locations (1):
- John D. Dingell VA Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No